CLINICAL TRIAL: NCT07097233
Title: The Impact of Virtual Reality Haptic Simulators and Mobile Apps on Manual Competence, Stress Levels, and Self-confidence of Dental Students in Endodontic Clinical Practice: A Randomized Clinical Trial
Brief Title: The Impact of Virtual Reality Haptic Simulators and Mobile Apps in Endodontic Clinical Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sıla Nur Usta, Professor (Associate), Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBU-GFOD-ENDO-SILANURUSTA-002
Record Dates: First submitted 2025-07-08; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Manual Dexterity; Self-Confidence; Stress Level
Keywords: dental education; dental students; educational virtual reality; endodontics; mobile app

STUDY DESIGN:
Intervention Model Description: Students will divided into 3 groups based on the received educational model before conducting endodontic treatment on real patients.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients who will be treated and the assessor who will assess the clinical scores of the students will be blinded regarding which educational method was used for the students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Haptic Simulator (Experimental): VRHS simulator will be used by dental students before treating a real patients in the endodontic clinical practice.
  Interventions: Procedure: Virtual Reality Haptic Simulator
- Mobile app (Experimental): Mobile app simulator will be used by dental students before treating a real patients in the endodontic clinical practice.
  Interventions: Procedure: Mobile app
- Control (Other): Control group will directly treat patients in the endodontic clinical practice withot prior exposure to any additional educational models
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Virtual Reality Haptic Simulator — Students will use a virtual reality haptic simulator as an adjunct educational tool before treating real patients in the clinical setting.
  Arms: Virtual Reality Haptic Simulator
Procedure: Mobile app — Students will use a mobile app as an adjunct educational tool before treating real patients in the clinical setting.
  Arms: Mobile app
Procedure: Control — Students will directly treat real patients without using virtual reality haptic simulator or mobile app.
  Arms: Control

SUMMARY:
Endodontics presents unique challenges due to the complexity and precision required in procedures such as access cavity preparation, canal instrumentation, and obturation. In this context, access cavity preparation is widely regarded as a critical step in endodontic treatment, as it facilitates the identification of the main root canal anatomy and enables effective chemomechanical debridement of the root canal system. However, the clinical application of this procedure can be particularly challenging for undergraduate students, as patients requiring endodontic care often present with varying degrees of anatomical complexity and clinical difficulty. These variations increase the of procedural complications. This is evident during the fourth year of dental education, when clinical endodontic training typically begins and students are required to perform their first treatments on patients. Initial attempts are often prone to failure due to limited theoretical knowledge, inadequate operative skills, and elevated stress levels. Therefore, ensuring comprehensive and well-structured preclinical training through the use of innovative educational strategies plays a critical role in both facilitating an effective transition to clinical practice and minimizing the risk of potential mishaps.The integration of virtual reality haptic simulators (VRHS) has shown considerable promise in enhancing the quality of endodontic preclinical education. VRHS provides students with an immersive, interactive environment that closely replicates real clinical scenarios, allowing for the development of tactile perception, fine motor control, and procedural accuracy in a risk-free setting. These simulators also encompass the potential drawbacks, such as a lack of standardized feedback and restricted opportunities for repetitive learning of traditional preclinical educational methods. In addition, through the advancements on the internet and mobile technology, mobile applications have become a game-changing tool for dental education. Mobile apps offer a flexible and self-paced learning environment that can be tailored to individual needs, thereby promoting greater engagement and a more interactive, immersive educational experience. As well as the VRHSs, mobile apps also simulate the clinical scenarios and procedures, providing students with the opportunity to develop and refine their skills within a structured and risk-free educational environment. Although the effectiveness of simulators has been investigated in endodontic preclinical settings using artificial teeth, their potential impact on real clinical performance and outcomes remains largely unexplored. Similarly, the role of mobile apps in endodontic education-particularly their effectiveness at the clinical level-has not been adequately studied.

DETAILED DESCRIPTION:
This three-arm randomized clinical study with an allocation ratio of 1:1:1 will be conducted in accordance with the Preferred Reporting Items for Randomized Trials in Endodontics (PRIRATE) 2020 guidelines. The study design was approved by the ethical committee of the University of Health Sciences (Approval No.: 2024-498). The sample size calculation was performed using G*Power 3.1.9.2 software, based on a significance level of 5% (α = 0.05), an effect size of 0.5997, and a statistical power of 80% (1-β = 0.80). The analysis indicated that a minimum of 10 students per group would be required to detect a statistically significant effect.

As part of the study, the VirTeaSy Dental simulator (VirTeaSy Dental©, France) will be utilized. This advanced system will feature an integrated touchscreen and a high-resolution three-dimensional (3D) display to provide detailed visualization of teeth, endodontic instruments, and clinical tools. Positioned beneath the 3D screen, haptic interfaces-including a dental mirror and a 3D mouse-will allow users to engage in a highly interactive and immersive simulation experience. Upon completion of each exercise, the simulator will generate a set of objective performance metrics, including surgery time (total procedure time in seconds), drilling time (duration of handpiece use in seconds), target progress (percentage of the intended area successfully removed), accuracy (percentage of non-targeted area preserved), target volume (volume of the intended area to be removed in mm³), and outside volume (volume of the area that should remain unaltered, in mm³).

As a mobile app, Dental EndoMaster (Dental-Edutec Inc., country) will be employed. This app will offer a unique, interactive 3D learning environment that simulates clinical scenarios using micro-CT-based models of teeth embedded within a virtual oral cavity. Users will be able to manipulate these models freely, with synchronized radiographic views and sectional visualizations that reveal internal anatomical structures. The app will include structured exercises guiding students through key procedures such as access cavity preparation and canal localization. Importantly, it will deliver real-time quantitative feedback on procedural metrics-including orifice estimation (%), adequate extension (%), overextension (%), and depth appropriateness (%)-enabling users to identify errors and monitor their performance.

All 4th-year dental students enrolled in the clinical endodontic training program will be invited to participate in the study. Prior to enrollment, the aims and scope of the study will be clearly communicated. Participants will be screened according to the following inclusion criteria: (1) having undergone similar training in access cavity preparation on extracted human teeth, with equivalent duration and methodology during their 2nd- and 3rd-year preclinical education from the same educator; (2) not having previous experience with the VRHS and/or mobile app; (3) having received the same theoretical lecture in endodontics; (4) not currently using medication for anxiety, depression, or systemic illness; (5) demonstrating at least a moderate level of computer literacy, as assessed by a standardized questionnaire; and (6) possessing baseline knowledge regarding access cavity preparation, determined by a brief theoretical quiz.

A total of 42 volunteer students will be anonymously assessed. Psychological distress and anxiety will be evaluated using the Patient Health Questionnaire-4 (PHQ-4) and the General Health Questionnaire-12 (GHQ-12). The PHQ-4, a validated four-item instrument, will be used to detect symptoms potentially impacting concentration and mood. The GHQ-12, a 12-item scale, will monitor variations in psychological distress throughout the study period. An online pre-evaluation test consisting of 10 multiple-choice questions on incisor access cavity preparation will be administered via the Kahoot platform (https://kahoot.it/), integrating gamification to enhance engagement. Students scoring ≥60 points will be eligible for inclusion. Computer literacy will be assessed using a modified self-assessment tool. Of the initial cohort, 30 students will meet the inclusion criteria and will be enrolled. Written informed consent will be obtained, and demographic data (age, gender) will be collected via a secure electronic form.

To maintain anonymity, each student will be assigned a randomized identification code. The 30 eligible students will be randomly assigned to three groups: Group 1 (VRHS, n=10), Group 2 (Mobile app, n=10), and Group 3 (Control, n=10). Prior to the study, the endodontists will hold a calibration meeting to review the study protocol and standardize instructional methods to minimize variability. All participants will receive a uniform introduction, including a live demonstration of access cavity preparation on maxillary incisors and a concise presentation on the VRHS and mobile apps, delivered by an experienced endodontist. Hands-on sessions will be conducted in small groups of five to promote engagement and ensure personalized supervision.

After the lecture and demonstration, students in Groups 1 and 2 will complete three practice sessions under standardized conditions to gain familiarity with the VRHS and mobile app, respectively. All sessions will be completed within one week, just before the students begin their clinical endodontic training. Following these sessions, a fourth trial will be performed using the respective technologies, during which performance metrics will be systematically recorded.

After completing the training phase, participants will proceed to perform access cavity preparations on randomly pre-assigned patients, following standardized clinical protocols under supervision. Group 3 students will perform clinical procedures without prior VRHS or mobile app training. Appointments will be scheduled to align with the beginning of the clinical internship. All patients will be informed about the study and will provide consent to be treated by students. Patient inclusion criteria will include: (1) ages 18-50 years, systemically healthy; (2) maxillary central/lateral incisors with apical periodontitis and only occlusal cavity; (3) absence of dental malformations; and (4) suitability for rubber dam isolation. Teeth with calcified canals, malformations, prosthetic preparation, prior endodontic treatment, or noncompliant patients will be excluded.

After completing their clinical sessions, students from all groups will perform the training sessions and fourth trial they had not previously experienced, and their respective performance metrics will be recorded.

Performance data from the fourth trial using the VRHS and mobile app will be automatically captured. The quality of clinical access cavity preparations will be assessed using a standardized assessment form, developed by expert endodontists. An independent and blinded evaluator will assess all clinical procedures and will record these as "clinical scores." Students will also perform self-evaluations using the same form, with these recorded as "self-clinical scores." This approach will allow comparison between expert evaluation and student-perceived performance. The clinical duration of access cavity preparation (in minutes) will also be documented.

Students' stress levels will be measured using a visual analog scale (VAS) at four stages: before initial use of VRHS or mobile app (VAS 0), after using the tools (VAS 1), immediately before (VAS 2), and immediately after clinical access preparation (VAS 3). Participants will complete a structured questionnaire to assess self-confidence and perceptions of the clinical training experience.

ELIGIBILITY:
Inclusion Criteria for dental students:

* having undergone similar training in access cavity preparation on extracted human teeth, with equivalent duration and methodology during their 2nd and 3th- years of preclinical education from the same educator
* not having previous experience regarding the use of VRHS and/or mobile app;
* having received the same theoretical lecture in endodontics
* not currently using any medication for anxiety, depression, or systemic illness
* demonstrating at least a moderate level of computer literacy, as assessed by a standardized questionnaire
* possessing a baseline knowledge regarding access cavity preparation, determined by a brief theoretical quiz.

Inclusion Criteria for included teeth:

* maxillary central or lateral incisors with apical periodontitis and only occlusal cavity
* teeth with absence of any dental malformations
* teeth suitable for rubber dam isolation.

Exclusion Criteria for dental students:

* Prior experience using virtual reality haptic simulators (VRHS) or the Dental EndoMaster mobile application
* Inconsistent or insufficient preclinical training in access cavity preparation (e.g., trained by a different educator, different duration or methodology).
* Did not attend or receive the same theoretical endodontics lecture as peers.
* Currently taking medications for anxiety, depression, or systemic illnesses that may affect cognitive or motor function.
* Demonstrating low computer literacy, as determined by a standardized self-assessment tool.
* Failing to achieve the minimum required score (e.g., <60 points) on the theoretical quiz about access cavity preparation.
* Refusal to provide informed consent or incomplete demographic/evaluation forms.
* Previous clinical experience in endodontics (e.g., performing real access cavity preparations on patients prior to the study).

Exclusion Criteria for teeth:

* Teeth other than maxillary central or lateral incisors (e.g., molars, premolars, mandibular teeth)
* Presence of extensive caries beyond occlusal cavity, restorations, or prosthetic crowns.
* History of previous endodontic treatment in the selected tooth.
* Dental malformations, such as dens invaginatus, dens evaginatus, or root anomalies.
* Calcified canals or limited canal visibility on radiographs
* Teeth not suitable for rubber dam isolation
* Patients with systemic diseases (e.g., immunocompromised, uncontrolled diabetes)
* Patients who are noncompliant, do not consent to student treatment, or express discomfort with participation in the study
* Pregnant or breastfeeding patients (optional, depending on ethical standards).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Manual dexterity | through study completion, an average of 1 day
  Measurements of clinical score and drilling time.
Stress | Baseline and through study completion, an average of 1 day
  Measurements of stress levels using VAS scale. This scale consists of a 10cm line, with two end points representing 0 ('no stress') and 10 ('stress as bad as it could possibly be').

SECONDARY OUTCOMES:
Self-confidence | through study completion, an average of 1 day
  Evaluation of the self confidence of students using a questionnaire that has been created by expert educators

IPD SHARING:
Plan to Share IPD: No
Within the scope of the necessity of protecting the individual information of the students and patients, it is considered that the recorded data will not be shared.

REFERENCES:
- [Background] Li Y, Ye H, Wu W, Li J, Zhao X, Liu Y, Zhou Y. Effectiveness and Methodologies of Virtual Reality Dental Simulators for Veneer Tooth Preparation Training: Randomized Controlled Trial. J Med Internet Res. 2025 May 22;27:e63961. doi: 10.2196/63961. PMID 40402564
- [Background] Patil S, Bhandi S, Awan KH, Licari FW, Di Blasio M, Ronsivalle V, Cicciu M, Minervini G. Effectiveness of haptic feedback devices in preclinical training of dental students-a systematic review. BMC Oral Health. 2023 Oct 10;23(1):739. doi: 10.1186/s12903-023-03410-3. PMID 37817151
- [Background] Suebnukarn S, Hataidechadusadee R, Suwannasri N, Suprasert N, Rhienmora P, Haddawy P. Access cavity preparation training using haptic virtual reality and microcomputed tomography tooth models. Int Endod J. 2011 Nov;44(11):983-9. doi: 10.1111/j.1365-2591.2011.01899.x. Epub 2011 May 28. PMID 21623838
- [Background] Bandiaky ON, Loison V, Volteau C, Cretin-Pirolli R, George S, Soueidan A, Le Guehennec L. Benefits of using immersive virtual reality in haptic dental simulation for endodontic access cavity training: A comparative crossover study. Int Endod J. 2025 May 12. doi: 10.1111/iej.14252. Online ahead of print. PMID 40353716
- [Background] Usta SN, Silva EJNL, Keskin C, Tekkanat H, Liukkonen M, Felszeghy S. A comparison of traditional and virtual reality haptic simulator approaches in preclinical endodontic training: Impacts on skill acquisition, confidence and stress. Int Endod J. 2025 Apr 10. doi: 10.1111/iej.14236. Online ahead of print. PMID 40207994